CLINICAL TRIAL: NCT05056090
Title: Effect of Prone Positioning on Mortality in Patients With Mild to Moderate Acute Respiratory Distress Syndrome.
Acronym: PROMILD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC20.366
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: ARDS; Acute Respiratory Distress Syndrome; Intensive Care Unit; Mechanical Ventilation
Keywords: ARDS; Acute Respiratory Distress Syndrome; Intensive Care Unit; ICU; Prone position
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: prospective, randomized, multicenter, open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will receive MV in PP (Experimental): Patients assigned to the intervention group will be turned in PP within the two hours after randomization for at least 16 consecutive hours. Then, patients will be turned in SP. Then, PP sessions are repeated as long as stopping criteria for PP are not met
  Interventions: Procedure: Patients will receive MV in PP
- Patients will receive MV in SP (No Intervention)

INTERVENTIONS:
Procedure: Patients will receive MV in PP — Putting the patient in a prone position
  Arms: Patients will receive MV in PP

SUMMARY:
Acute respiratory distress syndrome (ARDS) accounts for almost 10% of intensive care units (ICU) admissions. Three ARDS stages have been defined, based on the PaO2/FIO2 ratio measured with positive end-expiratory pressure (PEEP) ≥5 cmH2O: mild (201-300 mmHg), moderate (200-101 mmHg), and severe (≤100mmHg). They represent 30.0%, 46.6%, and 23.4% of ARDS, respectively.

Mechanical invasive ventilation (MV), the cornerstone of ARDS patient care, has a primary goal to protect the lung from ventilator-induced lung injury (VILI). Delivering MV in a prone position (PP) has been shown to improve oxygenation, protect the lung through a better homogenization of lung stress/strain, and stabilize hemodynamics.

A meta-analysis of four randomized controlled trials showed beneficial effect of PP vs. supine position (SP) in the most hypoxemic patients. A fifth randomized controlled trial further showed a significant reduction in mortality with PP in ARDS patients with PaO2/FIO2 <150 mmHg, when neuromuscular blockade and long prone positioning sessions were used. Therefore, PP has since been strongly recommended for ARDS patients with PaO2/FIO2 <150 mmHg. Yet, there is limited evidence in patients with mild to moderate ARDS.

There are, however, strong arguments supporting the need for a new trial in ARDS patients with PaO2/FIO2 in the range 150-300 mmHg:

1. There is no trial that has specifically tested PP in this ARDS subset;
2. PP is safe and has become a standard of care in ICU;
3. Should VILI prevention be a mechanism through which PP improves survival, this should be involved in all ARDS patients;
4. The mortality at hospital discharge in this subset of ARDS remains significant, amounting to 34.9% (95% confidence intervals 31.4-38.5%) in mild and 40.3% (37.4-43.3) in moderate stages;
5. Among 580 patients with mild ARDS at admission to the ICU, in-hospital mortality was 10%, 30%, and 37% for those who improved, persisted, and worsened ARDS, respectively.
6. Finally, PP has been shown to be cost-effective under commonly accepted thresholds.

The hypothesis is that in patients within the 150-300mmHg PaO2/FIO2 range at the time of ARDS diagnosis, PP can reduce mortality as compared to a similar group left in the SP.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or more admitted to ICU.
* ARDS patients meeting the Berlin criteria under invasive mechanical ventilation within the first 24h.
* Mechanically ventilated patients with standard settings: PEEP of 5 cmH2O or more and VT 6 ml/kg PBW and Pplat equal to or below 28-30 cmH2O after intubation.
* PaO2/FIO2 between 150 and 300 mmHg under previous settings within 12 hours after mechanical ventilation standardization.
* Written informed consent obtained from the patient, next of kin/proxy or emergency consent. The patient will be asked to give his consent for the continuation of the trial when his condition will allow.

Exclusion Criteria:

* Contra-indication to PP: spine instability; intracranial pressure greater than 20 mmHg; severe facial trauma; hemodynamic instability
* Non-inclusion criteria related to medical condition: Lung transplant; Burns over more than 20% of body surface; Chronic respiratory failure requiring home oxygen supplementation and/or non-invasive ventilation; Underlying disease with death expectancy within one year;
* Other non-inclusion criteria: Therapeutic limitation; inclusion into another interventional study in intubated and ventilated patients with mortality as primary end-point in the last 30 days; previously included in the same study; prone positioning before inclusion.
* Individuals referred to in Articles L. 1121-5 à L. 1121-7 (pregnant women, persons deprived of freedom, minors), adult individuals under protection of law (L. 1121-8 and L. 1122-1-2) (emergency situations) of public health regulation in France
* Patients not affiliated to social security insurance regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 28 days after inclusion
  All-cause mortality 28 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas TERZI, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France